CLINICAL TRIAL: NCT06537154
Title: Active Surveillance Versus Definitive Local Therapy for Patients Showing Clinical Complete Response Following Neoadjuvant Therapy for Muscle Invasive Bladder Cancer
Brief Title: NEO-BLAST: Neoadjuvant Therapy for Bladder Cancer Followed by Active Surveillance vs Treatment
Acronym: NEO-BLAST
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peter Black (Other)
Collaborators: University of British Columbia (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Peter Black, Professor, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H23-02447
Record Dates: First submitted 2024-07-29; First posted 2024-08-05 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Muscle-Invasive Bladder Carcinoma
Keywords: Muscle invasive bladder urothelial carcinoma; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Watchful Waiting; Circulating Tumor DNA; Magnetic Resonance Spectroscopy; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cCR, Standard of care (Active Comparator): Participants found to have a clinical complete response following NAT randomized to standard of care, described as "definitive bladder treatment", which consists of either radical cystectomy, or chemo-radiation of the bladder
  Interventions: Procedure: Control arm - Definitive bladder treatment
- cCR, Active surveillance (Experimental): Participants found to have a clinical complete response following NAT randomized to the investigational arm consisting of active surveillance. They will have have no local treatment to their bladder and will be monitored with cystoscopy, cytology and imaging (active surveillance)
  Interventions: Procedure: Active Surveillance
- non-cCR, standard of care (No Intervention): Participants found to have residual urothelial carcinoma (not cCR) will received the standard of care definitive bladder treatment. They will received either radical cystectomy or chemo-radiation of the bladder.

INTERVENTIONS:
Procedure: Active Surveillance — Participant found to have a cCR will be randomized to either standard of care or investigational active surveillance.
  Other Names: Clinical restaging (utDNA, ctDNA, MRI and TURBT)
  Arms: cCR, Active surveillance
Procedure: Control arm - Definitive bladder treatment — Standard of care, consisting of radical cystectomy or chemo-radiation of the bladder
  Arms: cCR, Standard of care

SUMMARY:
Invasive bladder cancer is managed with neoadjuvant therapy followed by bladder removal (cystectomy). Research shows that approximately 40% of patient will have no remaining cancer left in their bladder after completion of the initial systemic treatment, and perhaps could have avoided the surgery. However, currently physicians lack the ability to identify these patients.

The investigators believe that by using advanced imaging (MRI), bladder biopsies and novel biomarkers that detect tumor DNA in blood, they can better identify participants without any remaining cancer after chemotherapy. This will make active surveillance of these participants safer. In this study, participants without evidence of residual cancer will be randomized to active surveillance vs conventional bladder treatment (bladder removal, or chemo-radiation of the bladder). This study will be a pilot randomized control trial (RCT), and if successful, it will transition to a larger phase 3 RCT.

DETAILED DESCRIPTION:
Purpose To assess the feasibility to randomize patients with muscle-invasive bladder cancer (MIBC) who experience a complete clinical response (cCR) following neoadjuvant therapy (NAT), as defined by negative ctDNA, negative bladder MRI and negative repeat TURBT to active surveillance vs standard of care (SOC) with definitive bladder treatment.

Hypothesis The hypothesize is that the combination of bladder re-staging with MRI, repeat biopsy and the use of ctDNA will markedly enhance the ability to identified participant who achieve an excellent response to NAT (cCR) and who could safely be offered AS.

Justification:

Cisplatin-based neoadjuvant therapy (NAT) followed by radical cystectomy (RC), or alternatively in selected patient, a combination of chemo-radiation (trimodal therapy, TMT), are the current standards of care for treatment of MIBC. However, both have significant potential toxicity that can impact quality of life. Clinical trials have demonstrated that up to 38% of patients have a pathologic complete response (pCR) to NAT. Those patients could potentially avoid RC or TMT. Unfortunately, the clinical tools to predict pCR are still considered inadequate and definitive local therapy is advised. Retrospective data and now prospective phase 2 trials have reported promising outcomes in selected patients undergoing active surveillance. A prospective randomized trial is still lacking to ensure non-inferiority of active surveillance over the standard of care.

Primary Objectives:

* Phase 2 (pilot RCT): To determine the feasibility of randomizing patients with MIBC who experience a complete clinical response (cCR) following neoadjuvant treatment, as defined by negative ctDNA, negative bladder MRI and negative repeat TURBT, to active surveillance (AS) or definitive bladder treatment (DBT; consisting of radical cystectomy (RC) or trimodal therapy (TMT)).
* Phase 3: To estimate the metastasis-free survival rate at 2 years among patients with MIBC who experience a complete clinical response (cCR) following NAT, as defined by negative ctDNA, negative bladder MRI and negative repeat TURBT and who are managed with active surveillance.

Research design:

Multi-center, phase II/III, open label randomized clinical trial

After enrolment, participants will received SOC NAT. Blood and urine specimens will be collected before or at cycle 1 day 1 of NAT. Participants will undergo conventional restaging during NAT, recommended to be done at the end of cycle 2. Conventional imaging consists of computerized tomography (CT) scan of chest/abdomen/pelvis to rule-out local or distant progression on treatment. Participants who have successfully completed the full regimen of SOC NAT, and have not been found to have progression and/or metastasis on their SOC CT scan, will then undergo the following intervention for the "clinical restaging" (CRS) (must be completed within 4 weeks after last dose of NAT):

* ctDNA from blood samples collected before and after completion of NAT.
* Restaging bladder MRI
* Urine Cytology and Cystoscopy with template bladder biopsy under anesthesia with or without site-directed bladder biopsies.

Definition of clinical complete response (cCR):

* Absence of metastasis on conventional imaging.
* Negative MRI completed within 4 weeks of last dose of systemic treatment showing absence of VI-RADS 3, 4 or 5 lesion.
* Transurethral bladder tumor resection (TURBT) with or without site-directed bladder biopsies showing absence of high-grade carcinoma ≥cT1 and/or extensive and multifocal CIS. Focal CIS and/or completely resected Ta will be included in the definition of cCR and offered randomization.
* Negative ctDNA

Participants with cCR will then be randomized to either active surveillance or definitive bladder treatment (DBT) (RC or TMT, according to patient/physician choice). Participants who do not meet all criteria of cCR will proceed with SOC and have RC or TMT under the treating investigator's care.

Participants will adhere to the following schedule of surveillance:

Cystoscopy with urine cytology (for those with preserved bladder) every 3 months for 2 years. After 2 years, follow up schedule is at the discretion of the treating physician.

Repeat chest-abdomen-pelvis imaging with CT/MRI and ctDNA at 3, 6, 12, 18 and 24 months. After 2 years, follow up schedule is at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >18 years
* Primary urothelial or predominantly (>50%) urothelial carcinoma of the bladder with histologic evidence of muscularis propria invasion.
* Clinical stage T2-T4aN0M0 (Radiographic lymphadenopathy greater than 1.5 cm in short axis by imaging must be proven by biopsy to be free of cancer)
* No concomitant multifocal carcinoma in situ; a single focus is allowed.
* ECOG performance status 0, 1, or 2.
* Participants must be able to undergo pelvis MRI.
* Medically appropriate candidate for radical cystectomy (assessed by uro-oncologist) or chemo-radiation (assess by radiation-oncologist and medical-oncologist)
* Participants must be candidate to received standard of care (SOC) neoadjuvant systemic treatment at time of enrolment (assessed by medical-oncologist): 4 or more cycles of cisplatin-based chemotherapy (gemcitabine/cisplatin (GC) or methotrexate/vinblastine/Adriamycin/cisplatin (MVAC) or dose-dense MVAC (ddMVAC). If SOC evolves from the time of trial design and enrolment, eligibility to any SOC NAT (for example immunotherapy and/or antibody drug conjugate, as per NCCN guideline) will be allowed.
* Adequate bladder function and/or absence of significant urethral stricture to allow cystoscopic surveillance, as evaluate by urologist.

Exclusion Criteria:

* Any component of small cell or plasmacytoid histology.
* Prior systemic chemotherapy or immunotherapy (an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) or antibody-drug conjugate (NECTIN-4, HER2 or other) : Participants who have received any previous systemic therapy for urothelial carcinoma or cytotoxic chemotherapy, immunotherapy or other targeted therapy for another malignancy within 2 year of study entry are ineligible.
* No available bladder tumor tissue from prior TURBT for tumor sequencing.
* Prior or concurrent malignancy of any other site EXCEPT for non-melanoma skin cancer OR low risk malignancy not requiring treatment (such as prostate cancer Grade Group 1 under adequate surveillance, carcinoma in situ of the breast, cervix, etc.) AND unless free of disease for ≥ 5 years. Other cancers at low risk of recurrence may be allowed after review by principal investigator.
* Prior radiation therapy for bladder cancer.
* Participants who have received experimental agents within 4 weeks of study entry.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (defined by current oral or intravenous antibiotic therapy), symptomatic congestive heart failure (NYHA >2), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnancy. People of childbearing potential must have a negative serum pregnancy test before general anesthesia procedure and MRI
* No concurrent treatment on another clinical trial; supportive care trials or non-therapeutic trials (e.g., quality of life) are allowed.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders are eligible
Enrollment: 688 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients found to have a cCR and randomized on the number of patients enrolled (pilot-RCT ; phase 2) | 24 months
  Feasibility to randomized patients with cCR to either active surveillance or definitive bladder treatment.
Metastasis free survival at 2 years (phase 3) | 24 months
  Time to metastasis, defined as >cN1 (more than 1 clinically suspicious lymph nodes), cT4a (unresectable disease), or M1 disease or death.

SECONDARY OUTCOMES:
Bladder-intact event-free survival | 24 months
  Time from study entry to the earliest of histologically proven presence of MIBC (≥T2), clinical evidence of nodal or metastatic disease, radical cystectomy, or death due to any cause.
Proportion of cCR patient with ypT0 | 24 months
  Rate of ypT0 (pathologic complete response) on cystectomy specimen following NAT in participants who had a cystectomy after identification of cCR.
Overall survival | 24 months
  Time from study entry to death; individuals who are alive at last contact will be censored on the date of last contact.
Acceptance rate to treatment allocation | 6 months
  Rate of concordance between treatment allocated and treatment received within the first 3 months following randomization.
Quality of life measure by EORTC-QLQ-C30 in participants according to treatment received | 24 months
  European Organisation for Research and Treatment of Cancer QLG Core Questionnaire (EORTC QLQ-C30). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher (better) response level and quality of life.
Quality of life measure by EORTC QLQ BLM-30 in participants according to treatment received | 24 months
  European Organisation for Research and Treatment of Cancer - Muscle-Invasive Bladder Cancer Module 30 (EORTC QLQ BLM-30). All of the Multi-item scales and Single-item measures range in score from 0 to 100. A high score for all of the Multi-item scales excluding Sexual functioning, and for the Single item, represents a high level of symptomatology or problems (worse outcome), whereas a high score for the Sexual functioning scale represents a high level of functioning (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Black, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Prostate Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared publicly. The decision to not share IPD is based on considerations regarding participant privacy and confidentiality. However, data sharing may be considered on a case-by-case basis upon request and subject to approval by the Principal Investigator. Interested researchers can direct inquiries to the Principal Investigator, and each request will be evaluated to ensure compliance with participant privacy and confidentiality policies. Aggregate data and study results will be shared through publications and presentations.